CLINICAL TRIAL: NCT00888771
Title: Characterisation of Small Colonic Polyps in Vivo
Brief Title: Discard:Characterisation of Colonic Polyps in Vivo
Acronym: DISCARD
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 05/Q0405/121/1
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Polyps
Keywords: Colorectal cancer; polyps; colonoscopy; advanced imaging
MeSH Terms: conditions — Colorectal Neoplasms; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1
- 2
- 3
- 4

SUMMARY:
Prospective study of accuracy of colonic polyp characterisation in vivo using high resolution white light endoscopy, narrow band imaging and chromoendoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age, assessed as fit for routine colonoscopy
2. Patients attending for screening or surveillance colonoscopy meeting the following criteria:

   * Polyp surveillance with at least 3 adenomas or 1 adenoma>10mm at previous colonoscopy
   * Surveillance post colorectal cancer resection
   * Screening with positive faecal occult blood test

Exclusion Criteria:

1. Patients with known colitis or polyposis syndromes
2. Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group therefore would comprise those presenting for 3 yearly follow up or sooner i.e. those with a resected colorectal cancer or those with ≥ three adenomas or one advanced ≥10mm adenoma or those with a positive faecal occult blood test
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of polyp characterisation | 12 months

SECONDARY OUTCOMES:
Change in surveillance interval after formal histopathology | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Saunders, MD, Principal Investigator — Wolfson Unit for Endoscopy, St Mark's Hospital
Locations (1):
- Wolfson Unit for Endoscopy, St Mark's Hospital, Harrow, Moddlesex, United Kingdom

REFERENCES:
- [Derived] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250